CLINICAL TRIAL: NCT02750813
Title: ACUVUE® OASYS® 1-DAY vs DAILIES TOTAL1®: Clinical Comparison in a Symptomatic Population
Brief Title: ACUVUE® OASYS® 1-DAY vs DAILIES TOTAL1®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon, a Novartis Company (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLV771-P001
Record Dates: First submitted 2016-04-21; First posted 2016-04-26 (Estimated); Results first posted 2017-09-26 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-08

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DT1, then AO1D (Other): Delefilcon A contact lenses worn first, followed by senofilcon A contact lenses. Each product worn bilaterally (in both eyes) for 14 days in a daily wear, daily disposable modality.
  Interventions: Device: Delefilcon A contact lenses; Device: Senofilcon A contact lenses
- AO1D, then DT1 (Other): Senofilcon A contact lenses worn first, followed by delefilcon A contact lenses. Each product worn bilaterally for 14 days in a daily wear, daily disposable modality.
  Interventions: Device: Delefilcon A contact lenses; Device: Senofilcon A contact lenses

INTERVENTIONS:
Device: Delefilcon A contact lenses
  Other Names: DAILIES TOTAL1® (DT1)
Device: Senofilcon A contact lenses
  Other Names: ACUVUE® OASYS 1-Day with HydraLuxe™ (AO1D)

SUMMARY:
The purpose of this study is to compare the lens fit characteristics, specifically lens centration, of ACUVUE® OASYS® 1-DAY (AO1D) contact lenses and DAILIES TOTAL1® (DT1) contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Must sign informed consent form;
* Adapted, current daily disposable soft contact lens wearer who typically wears lenses every day, or at least 5 days per week, 6 hours per day;
* Symptoms of contact lens discomfort as defined by the Symptomatology (Eligibility) Pre-screening questionnaire;
* Prescription within -1.00 Diopter (D) to -6.00D to be fitted with study contact lenses;
* Cylinder equal or lower than -0.75D in both eyes;
* Vision correctable to 20/25 or 0.1 logMAR (Logarithmic minimum angle of resolution) or better in each eye at distance with both study lenses at Visit 1;
* Can be successfully fitted with both study lenses at Visit 1;
* Willing to wear lenses every day or at least 5 days per week, 6 hours per day and attend all study visits;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Ocular anterior segment infection, inflammation, abnormality, or active disease that would contraindicate contact lens wear;
* Use of systemic or ocular medications for which contact lens wear could be contraindicated as determined by the Investigator;
* Monocular (only 1 eye with functional vision) or fit with only 1 lens;
* Fitted with monovision;
* Prior refractive surgery;
* History of herpetic keratitis, ocular surgery, or irregular cornea;
* Pregnant or lactating;
* Use of mechanical eyelid therapy or eyelid scrubs within 14 days before Visit 1 and not willing to discontinue during the study;
* Participation in any clinical study within 30 days of Visit 1;
* Current DT1 or AO1D lens wearer;
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2016-08-17 (Actual); Study Completion 2016-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Manager, Global Medical Affairs, GCRA, Study Director — Alcon, A Novartis Division
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 12 study centers located in the United States.
Pre-assignment Details: Of the 252 enrolled, 5 subjects were exited prior to randomization and 1 randomized subject was exited prior to treatment. This reporting group includes all randomized subjects who were exposed to a study product (test or control) (246).
Period: Period 1, First 14 Days of Wear
Arm/Group | DT1, Then AO1D | AO1D, Then DT1
Started | 125 | 121
Completed | 124 | 120
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Reason not given | 0 | 1
Period: Period 2, Second 14 Days of Wear
Arm/Group | DT1, Then AO1D | AO1D, Then DT1
Started | 124 | 120
Completed | 124 | 120
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects who were exposed to any study lens, except for lenses used at Visit 1 for parameter optimization and fitting (Full Analysis Set).
Groups:
- Overall: Delefilcon A and senofilcon A contact lenses worn during Period 1 and Period 2 in a crossover assignment.
Arm/Group | Overall
Number analyzed (Participants) | 246
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (8.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183
  Male | 63

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Lenses Graded as 0 or 1 for Lens Centration at Day 14
Description: Lens centration, was assessed by the investigator for each eye individually and rated on a 5-point scale: 0=centered/optimal, 1=slight decentration, 2=mild decentration, 3=moderate decentration, 4=severe decentration. The combined percentage of lenses assessed as "centered" or "slight decentration" is reported. Lenses from both eyes contributed to the percentage.
Time Frame: Day 14, each product
Population: Full Analysis Set. Number Analyzed is the number of eyes with non-missing response.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: Eyes
Groups:
- DAILIES TOTAL1: Delefilcon A contact lenses worn bilaterally for 14 days in a daily wear, daily disposable modality
- AO1D: Senofilcon A contact lenses worn bilaterally for 14 days in a daily wear, daily disposable modality
Arm/Group | DAILIES TOTAL1 | AO1D
Number analyzed (Participants) | 244 | 244
Number analyzed (Eyes) | 488 | 488
percentage of lenses | 100.0 | 99.4

2. Secondary Outcome: Ex Vivo Critical Coefficient of Friction (CCOF) at Day 14
Description: The ex vivo CCOF (ratio of the force of friction between two bodies and the force pressing them together) was measured by the incline plane technique after 16 hours of lens wear. Worn lenses were collected and analyzed for a subset of subjects (all subjects from one site only) who attended the Day 14 visit (Visit 2 and Visit 3) after 16 hours of lens wear. Only lens worn on the right eye (OD) was measured in each subject per each lens brand. CCOF values for contact lenses range from near zero to approximately 0.10 using the inclined plane method. A lower CCOF indicates higher contact lens lubricity.
Time Frame: Day 14, each product
Population: Full Analysis Set. Number Analyzed is the number of eyes with non-missing responses, including only subjects from one site.
Measure: Mean (Standard Deviation); unit: unitless
Units Other Than Participants: Eyes
Arm/Group | DAILIES TOTAL1 | AO1D
Number analyzed (Participants) | 17 | 17
Number analyzed (Eyes) | 17 | 17
unitless | 0.0468 (0.00557) | 0.0675 (0.00599)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent for the duration of a subject's participation in the study (up to 35 days). AEs are reported as pre-treatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the medical device.
Groups:
- Pretreatment: All subjects who consented to participate in the study prior to initiation of study treatment
- DAILIES TOTAL1 (DT1): All subjects exposed to DT1 contact lenses, except for lenses used for parameter optimization and fitting
- ACUVUE OASYS 1-DAY (AO1D): All subjects exposed to AO1D contact lenses, except for lenses used for parameter optimization and fitting
Arm/Group | Pretreatment | DAILIES TOTAL1 (DT1) | ACUVUE OASYS 1-DAY (AO1D)
All-Cause Mortality (participants affected / at risk) | 0/252 | 0/246 | 0/246
Serious Adverse Events (participants affected / at risk) | 0/252 | 0/246 | 0/246
Other Adverse Events (participants affected / at risk) | 0/252 | 0/246 | 0/246

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.